CLINICAL TRIAL: NCT04509232
Title: "Parental Perception and Acceptance of the Utilization of Silver Diamine Fluoride on Their Child's Anterior and Posterior Teeth Before and After Masking the Colour With Glass Ionomer"
Brief Title: Assessing Parental Acceptance to Silver Diamine Fluoride Staining Before and After Masking the Colour With Glass Ionomer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dina Bassam Mohamed Ahmed (Other)
Responsible Party: Sponsor-Investigator, Dina Bassam Mohamed Ahmed, Dina Bassam Mohamed Ahmed, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PED1931M
Record Dates: First submitted 2020-08-08; First posted 2020-08-11 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Caries Arrested
Keywords: Tertiary prevention; Remineralizing agent
MeSH Terms: interventions — silver diamine fluoride; glass ionomer

STUDY DESIGN:
Intervention Model Description: Involves two groups of participants. One group receives
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): - 38% Silver diamine fluoride will be applied to carious lesions by microbrush on the affected surface application time should be 1 min, Application time will be shorter in very young patients.
  Interventions: Procedure: Silver diamine fluoride
- group B (Experimental): -38% Silver diamine fluoride will be applied by the same protocol as in group A
  Then Glass Ionomer restoration is applied as follows
  * Self cure glass ionomer restoration is applied not light cured as light causes oxidation of silver and the filling appears darker.
  * Glass ionomer won't be applied immediately after SDF placement it will be applied at time ranging from 2 hours to two days.
  * Conditioning of the base of the cavity is done by 3M ESPE conditioner for 10 seconds then rinsing the cavity for 10 to 20 secs.
  * Applying High strength hand mix chemical self cure glass ionomer.
  Interventions: Procedure: Silver diamine fluoride and glass ionomer

INTERVENTIONS:
Procedure: Silver diamine fluoride — Group A
  * Excavation of soft carious dentin will be done to minimize the staining.
  * The selected teeth should be cleaned, dried and isolated. Vaselline should be applied to surrounding soft tissues to avoid their staining.-
  * 38% Silver diamine fluoride will be applied to carious lesions by microbrush
  * Apply gentle flow of air until medicament is dry, Try to keep isolated for three minutes,remove excess SDF with cotton pellet to decrease systemic absorption.
  After silver diamine fluoride application Assessement of parental acceptance to staining will be done though a 5 point likert scale For anterior and posterior teeth separately .
  Other Names: SDF
  Arms: group A
Procedure: Silver diamine fluoride and glass ionomer — * 38% Silver diamine fluoride will be applied by the same protocol as in group A Then Glass Ionomer restoration is applied
  * Parental acceptance to staining will be assessed thought 5 point likert scale after application of SDF and once more after application of Glass Ionomer restoration.
  Other Names: SDF; GIC
  Arms: group B

SUMMARY:
Assessing Parents acceptance for the colour of Silver Diamine Fluoride on their Children anterior and posterior teeth before and after masking its colour with Glass Ionomer.

DETAILED DESCRIPTION:
Sample size estimation Sample size estimation was based on the primary outcome of interest The final sample size was 41 children per group (total sample size = 82 children)

Patients will be recruited randomly from outpatient clinic of the Department of Pediatric Dentistry and Dental Public Health, Faculty of Dentistry, Ain Shams University. A signed informed consent to the parents' and also an insent to child,outlined by the Ethical Committee, Faculty of Dentistry, Ain Shams University will be obtained before the conduction of the study.

All examination procedures will be done by the same operator to ensure standardization.

Moreover, all patients will receive oral health education in regard to dietary and oral hygiene habits.

Excluded carious primary molars will be scheduled to receive the appropriate treatment.

Before applying any procedures medical history for any silver products allergy (SDF allergy) will be assessed by asking the child's parent.

Materials:

38%SDF

Conditioner 3M ESPE

High strength hand mix chemical cure glass ionomer

Patient withdrawal

Patient who don't comply to the oral hygiene given will be excluded from the study.

Patients who are not willing to continue in the study will have the right to quit at any time without loss of any benefits.

Data Management

Patient information will be gathered and stored in the patient examination chart of the outpatient clinic, Department of Pediatric Dentistry, faculty of Dentistry, Ain Shams University.

All information will be kept as a hard copy and as an electronic one as well. Patient information will be guarded as confidential information that should never be revealed at all times.

Adverse Event Reporting

SDF is not expected to have any adverse effects on healthy subjects, yet failure of treatment, recurrent caries, abcess formation or pulpal affection may be an issue of concern, that will be avoided by the continuous follow up sessions.

Statistical Analysis

Sample size estimation was based on the primary outcome of interest, which is to test whether there's a significant difference in parent satisfaction between the parents of children receiving SDF and those receiving SDF followed by ART restorations. The predicted sample size for comparing parent satisfaction score was found to be 34 children per group (total sample size = 68 children), by assuming an α level of 0.05 and β level of 0.2 (power = 80%). The effect size d was calculated based on the findings of M. Jiang, et al., and the allocation ratio was set at 1. After adjusting for 20% dropout, the final sample size was 41 children per group (total sample size = 82 children). Sample size calculation was performed using G*Power software version 3.1.4 for MS Windows.

ELIGIBILITY:
Inclusion Criteria:

1. Uncooperative patients.
2. Patients whom their parents refuse or cannot afford the cost of GA surgeries.
3. Teeth that are restorable with restoration and doesn't need full coverage.
4. Teeth which are free of symptoms of pulpal pathology.
5. Children with anterior and posterior carious teeth with minimum of two teeth.

Exclusion Criteria:

1. Patients whom their parents totally refuse Silver diamine fluoride staining .
2. Children suffering from any medical condition that can't be managed in the clinic.
3. Children with known allergies to silver products.
4. Children with severe forms of hypoplasia .

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 82 (Actual)
Dates: Start 2019-10-12 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-09-22 (Actual)

PRIMARY OUTCOMES:
Assessement of Parental perception and Acceptance | december 2019 to june 2021
  Assessement of Parental Perception and Acceptance of the Utilization of Silver Diamine Fluoride on their Child's Anterior and Posterior Teeth before and after masking the colour with Glass Ionomer through 5 point likert scale
  The format of the five-level Likert scale will be
  1. Strongly disagree
  2. Disagree
  3. Neutral
  4. Agree
  5. Strongly agree

SECONDARY OUTCOMES:
protocol for placement of silver diamine fluoride with minimal staining | december 2019 to june 2021
  Applying a protocol for placement of silver diamine fluoride with minimal staining as an alternative modality to general anesthesia for treatment of uncooperative patients in the department of pediatric dentistry Ain shams university.

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anil S, Anand PS. Early Childhood Caries: Prevalence, Risk Factors, and Prevention. Front Pediatr. 2017 Jul 18;5:157. doi: 10.3389/fped.2017.00157. eCollection 2017. PMID 28770188
- [Background] Clemens J, Gold J, Chaffin J. Effect and acceptance of silver diamine fluoride treatment on dental caries in primary teeth. J Public Health Dent. 2018 Dec;78(1):63-68. doi: 10.1111/jphd.12241. Epub 2017 Jul 27. PMID 28749529
- [Background] Innes NP, Manton DJ. Minimum intervention children's dentistry - the starting point for a lifetime of oral health. Br Dent J. 2017 Aug 11;223(3):205-213. doi: 10.1038/sj.bdj.2017.671. PMID 28798464
- [Background] Caries-risk Assessment and Management for Infants, Children, and Adolescents. Pediatr Dent. 2018 Oct 15;40(6):205-212. No abstract available. PMID 32074889
- [Background] Zhao IS, Gao SS, Hiraishi N, Burrow MF, Duangthip D, Mei ML, Lo EC, Chu CH. Mechanisms of silver diamine fluoride on arresting caries: a literature review. Int Dent J. 2018 Apr;68(2):67-76. doi: 10.1111/idj.12320. Epub 2017 May 21. PMID 28542863
- [Background] JUCSF protocol for caries arrest using silver diamine fluoride: rationale, indications, and consent. Br Dent J. 2017 Apr 7;222(7):516. doi: 10.1038/sj.bdj.2017.311. PMID 28387277
- [Background] Policy on the Use of Silver Diamine Fluoride for Pediatric Dental Patients. Pediatr Dent. 2018 Oct 15;40(6):51-54. No abstract available. PMID 32074849
- [Background] Crystal YO, Niederman R. Evidence-Based Dentistry Update on Silver Diamine Fluoride. Dent Clin North Am. 2019 Jan;63(1):45-68. doi: 10.1016/j.cden.2018.08.011. PMID 30447792
- [Background] Burgess JO, Vaghela PM. Silver Diamine Fluoride: A Successful Anticarious Solution with Limits. Adv Dent Res. 2018 Feb;29(1):131-134. doi: 10.1177/0022034517740123. PMID 29355424
- [Background] Crystal YO, Janal MN, Hamilton DS, Niederman R. Parental perceptions and acceptance of silver diamine fluoride staining. J Am Dent Assoc. 2017 Jul;148(7):510-518.e4. doi: 10.1016/j.adaj.2017.03.013. Epub 2017 Apr 27. PMID 28457477
- [Background] Chu CH, Lee AH, Zheng L, Mei ML, Chan GC. Arresting rampant dental caries with silver diamine fluoride in a young teenager suffering from chronic oral graft versus host disease post-bone marrow transplantation: a case report. BMC Res Notes. 2014 Jan 3;7:3. doi: 10.1186/1756-0500-7-3. PMID 24383434
- [Background] Alshammari AF, Almuqrin AA, Aldakhil AM, Alshammari BH, Lopez JNJ. Parental perceptions and acceptance of silver diamine fluoride treatment in Kingdom of Saudi Arabia. Int J Health Sci (Qassim). 2019 Mar-Apr;13(2):25-29. PMID 30983942